CLINICAL TRIAL: NCT05416866
Title: Transversus Abdominis Plane Block Plus Quadratus Lumborum Block or Retrolaminar Block of Multiple Injections for Postoperative Analgesia Following Laparoscopic Colorectal Surgery: A Randomized, Double-blind, Controlled Trial
Brief Title: Transversus Abdominis Plane Block Plus Quadratus Lumborum Block or Retrolaminar Block of Multiple Injections for Postoperative Analgesia Following Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: dong zhang (Other)
Responsible Party: Sponsor-Investigator, dong zhang, Anesthesiologist, Gansu Provincial Hospital
Organization: Gansu Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GanSu Province
Record Dates: First submitted 2022-05-26; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Quadratus Lumborum Block; Analgesia; Laparoscopic; Colorectal
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Except the regional anesthesiologist who performed the blocks, patients, surgeons, theatre anesthesiologists, ward staff, caregivers, and the outcome assessor were unaware of group allocation. The regional anesthesiologist was not involved in the other parts of the study. All data was collected by personnel blinded to the patient group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TR group (Experimental): ultrasound-guided transversus abdominis plane block with 20 ml mixture 0.20% ropivacaine + dexamethasone 5 mg and retrolaminar block with 30-40 ml mixture 0.20% ropivacaine + dexamethasone 5 mg
  Interventions: Procedure: Retrolaminar block on the operative side; Procedure: Transversus abdominis plane block on the nonoperative side
- TQ group (Experimental): ultrasound-guided transversus abdominis plane block with 20 ml mixture 0.20% ropivacaine + dexamethasone 5 mg and quadratus lumborum block with 30 ml mixture 0.20% ropivacaine + dexamethasone 5 mg
  Interventions: Procedure: Quadratus lumborum block on the operative side; Procedure: Transversus abdominis plane block on the nonoperative side

INTERVENTIONS:
Procedure: Retrolaminar block on the operative side — After the skin near the puncture site was disinfected, 2ml of 1% lidocaine was injected into the puncture site for local infiltration. The needle was inserted beneath the ultrasound probe using an in-plane orientation to contact the lamina of the T8-T11 vertebra. Then we retracted the tip of needle to the lamina about 1 mm and withdrew to make sure that there was no blood or cerebrospinal fluid. Then, 30-40 mL mixture was injected posterior to the lamina of T8-T11.
  Arms: TR group
Procedure: Quadratus lumborum block on the operative side — In our study, we applied a transmuscular approach to the QLB. After the patients were placed in the lateral position, the skin near the puncture site was disinfected, a low-frequency (3-5 MHz), curvilinear probe is used and is located vertical to the iliac crest at the posterior axillary line to find the Shamrock sign. After the local infiltration for puncture site, the 22-G needle is then inserted in plane and directed to the QL muscle. After the proper position of the needle tip between the psoas major muscle and the QL muscle is confirmed, 30 ml mixture is injected into the interfascial plane.
  Arms: TQ group
Procedure: Transversus abdominis plane block on the nonoperative side — After placing the patients in the supine position, the skin was disinfected. A linear probe was placed in the transverse plane at the midaxillary line between the lower costal margin and iliac crest. When the external oblique, internal oblique, and transversus abdominis muscles were observed, 2ml of 1% lidocaine was injected into the puncture site for local infiltration.Then, a 22-gauge, 80-mm needle was advanced using an in-plane technique in an anteromedial to posterolateral direction toward the TAP (the fascial plane between the internal oblique and transversus abdominis muscles). After the correct position of the needle tip was verified, 20 ml mixture was injected into the TAP. The ultrasound showed that the local anesthetic separated the internal oblique and transversus abdominis muscles, confirming the success of the block.

SUMMARY:
Our hypothesis was that transversus abdominis plane block plus retrolaminar block would reduce postoperative sufentanil consumption and provide superior analgesia compared with transversus abdominis plane block plus quadratus lumborum block for laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II class
* Colorectal cancer patients
* 18 and 80 years old
* Elective laparoscopic colorectal surgery

Exclusion Criteria:

* serious complications associated with other systems:
* severe cardiac insufficiency
* renal failure
* hepatic encephalopathy
* infection in the block injection area
* coagulopathy
* a known allergy to local anesthetics
* a previous history of tranquilizer or opioid abuse,
* body mass index (BMI) greater than 30 kg/m2 or less than 18 kg/m2,
* inability to cooperate with the assessment of visual analogue scale (VAS) pain scores
* refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
the cumulative consumption of sufentanil | 24 hours after nerves block
  the outcome in micrograms

SECONDARY OUTCOMES:
the patient's mean arterial pressure (MAP), HR at rest and during movement at 1, 2, 4, 6, 8, 12, 18, 24 after nerves block | the time for completion of nerves block was time 0
  MAP in mmHg, HR in rate/one minute.
cumulative sufentanil consumption at predetermined time intervals | within 24 hour after nerves block
  the outcome in minutes
time until the earliest single patient-controlled analgesia (PCA) dose of sufentanil | within 24 hour after nerves block
  the outcome in minutes
the number of PCA press | within 24 hour after nerves block
  the outcome in frequency
time until the earliest rescue analgesia and antiemetic | within 24 hour after nerves block
  the outcome in minutes
the total dose of rescue analgesia and antiemetic | within 24 hour after nerves block
  the outcome in milligrams
block-related complications | within 24 hour after nerves block
  such as hematoma, infection, quadriceps weakness, pneumothorax, deep visceral injury, and evidence of systemic toxicity to the local anesthetic
other side events | within 24 hour after nerves block
  such as bradycardia (HR less than 60 beats per min), hypotension (systolic blood pressure less than 90 mmHg or more than 20% lower than baseline), hypoxemia (SpO2 less than 90%), respiratory depression (RR less than 10 breaths per min lasting for more than 10 min), pruritus, backache, nausea and vomiting
patient satisfaction with pain management | at 24th hour after nerves block
  Patient satisfaction on postoperative analgesia using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied, and 5 = very satisfied)
the length of hospital stay | up to 2 weeks
  the outcome in days
Visual Analog Score (VAS) for pain at rest and during movement at 1, 2, 4, 6, 8, 12, 18, 24 after nerves block | the time for completion of nerves block was time 0
  The VAS is an internationally recognized scale for assessment of pain on an 11-point scale ranging from 0 to 10 points, with 0 defined as no pain and 10 defined as the worst pain imaginable (units on a scale)